CLINICAL TRIAL: NCT06474052
Title: Volume Kinetics of Gelofusine 4% During Uncomplicated Vascular Surgery
Brief Title: Volume Kinetics of Gelofusine 4% During Vascular Surgery
Status: Completed | Type: Observational
Sponsor: Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu (Other)
Responsible Party: Principal Investigator, Balan Ion Cosmin, Principal Investigator, Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu
Other Study IDs: 1391
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Fluid Electrolyte Disorders
Keywords: colloid; volume kinetics; Gelofusine 4%
MeSH Terms: interventions — Colloids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Gelofusine 4%: Adult patients undergoing uncomplicated vascular surgery.
  Interventions: Drug: Gelofusine 4%

INTERVENTIONS:
Drug: Gelofusine 4% — Gelofusine 4% 10 ml/kg is administered following anaesthesia induction in 30 minutes.
  Other Names: Colloid

SUMMARY:
The volume kinetics of the commercially available colloid fluid, Gelofusine 4%, have not been previously studied. Adult patients undergoing open vascular surgery, including femoral and carotid endarterectomy as well as bypass surgery, received general anesthesia. Following the induction of anesthesia, Gelofusine 4% was administered at a dosage of 10 ml/kg over a 30-minute period. Hemoglobin concentration was monitored for up to 180 minutes post-administration to construct a plasma hemodilution profile.

DETAILED DESCRIPTION:
Gelofusine 4% was administered at a dosage of 10 ml/kg over a 30-minute period to adult patients undergoing uncomplicated vascular surgery. Arterial blood samples were taken to measure blood hemoglobin concentration and hematocrit at baseline and at 5-minute intervals up to 60 minutes after the infusion began, followed by 10-minute intervals up to 90 minutes, and then at 30-minute intervals up to 180 minutes. Urine output and total intraoperative blood loss were continuously monitored. The plasma hemodilution data were fitted to a bicompartmental model to derive the intercompartmental kinetics of Gelofusine 4%.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Elective open vascular surgery with a minimal risk of perioperative complications.
* Hemodynamic stability before induction (no chest pain, SBP > 100 mmHg, MAP ≥ 60 mmHg, 50 < HR < 100 bpm).

Exclusion Criteria:

* Known allergy to 4% Gelofusine.
* Patient refusal to participate in the study.
* Non-elective/emergency surgical interventions.
* The American Society of Anesthesiologists (ASA) > 3.
* Any preoperative hemodynamic support (mechanical or pharmacological).
* Moderate or severe left ventricular dysfunction (LVEF ≤ 44%).
* Moderate or severe right ventricular dysfunction.
* Diastolic dysfunction of any degree.
* Baseline hypoxemia index < 300 mmHg.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 80 years undergoing uncomplicated vascular surgery under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Plasma Volume | 180 minutes after the start of the Gelofusine 4% infusion
  Plasma volume was determined using a two-compartment kinetic model with three rate constants (k12, k21, and k10) and a scaling factor (Vc, central volume) that relates dilution to volume. This model was applied to the dependent variables, which included frequently measured plasma dilution and urinary excretion.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hahn, Professor, Study Director — Karolinska Institutet: Stockholm, SE (Department of Clinical Sciences, Danderyd Hospital) Employment
Locations (1):
- Institutul de Urgenta de Boli Cardiovasculare Prof Dr CC Iliescu, Bucharest, București, Romania

REFERENCES:
- [Derived] Balan C, Boros C, Bubenek-Turconi SI, Hahn RG. Volume Kinetics of Gelofusine 4% During Vascular Surgery. Clin Pharmacokinet. 2025 Apr;64(4):599-610. doi: 10.1007/s40262-025-01500-9. Epub 2025 Mar 23. PMID 40121598